CLINICAL TRIAL: NCT04589949
Title: Early Convalescent Plasma Therapy for High-risk Patients With COVID-19 in Primary Care (the CoV-Early Study)
Acronym: CoV-Early
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: vaccination uptake 80% in the target population/new COVID variant
Sponsor: Erasmus Medical Center (Other)
Collaborators: Prothya Biosolutions (Industry); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Bart Rijnders, MD, PhD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL74972.078.20
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ConvP (Experimental): 300 mL convalescent plasma with a minimum of neutralizing antibodies
  Interventions: Biological: ConvP
- FFP (Active Comparator): 300 mL Fresh Frozen plasma
  Interventions: Biological: FFP

INTERVENTIONS:
Biological: ConvP — Infusion of plasma retrieved from donors with a history of PCR proven symptomatic COVID.
  Plasma will be administered according to the Erasmus MC KIS protocol regarding the use of blood products
  Other Names: convalescent plasma
  Arms: ConvP
Biological: FFP — Infusion of thawed non-convalescent plasma Plasma will be administered according to the Erasmus Medical Center quality protocol regarding the use of blood products
  Other Names: Fresh Frozen Plasma
  Arms: FFP

SUMMARY:
An effective, widely available, and safe treatment that can decrease the duration, severity and fatality of COVID-19 is urgently needed. Also, in the most affected regions the pressure on health care systems including ventilator support capacity can be a limiting factor for survival. Initial studies including from our group indicate that administering convalescent plasma containing high titers of neutralizing antibodies to COVID-19 patients who are already relatively late during the disease course after hospital admission is not effective, which can be explained by high titers of autologous antibodies present in patients. Thus, the antiviral capacity of convalescent plasma is hypothesized to be best positioned early in the disease course and in patients at increased risk for a severe disease course. If effective, any treatment that decreases the need for hospital admission is very valuable but so far, no COVID-19 treatment has been shown to prevent clinical deterioration when given before patients are admitted to the hospital.

Primary objective:

To evaluate the efficacy, feasibility and safety following the administration of convalescent plasma (ConvP) as a therapy for outpatients diagnosed with COVID-19 at increased risk for an unfavourable clinical outcome and within 7 days after symptom onset.

Study design:

This trial is a nationwide multicenter, double blind, randomized controlled trial in the Netherlands. Patients will be randomized between the transfusion of 300mL of convP versus regular fresh frozen plasma (FFP).

Patient population:

Patients with polymerase chain reaction (PCR) confirmed COVID disease with less than 8 days of symptoms, age 70 or older or 50-69 years with at least 1 additional risk factor for severe COVID-19 are eligible.

Intervention:

300mL of convP with a minimum level of neutralizing antibodies.

A total of 690 patients will be included. Expected duration of accrual: 18-24 months Duration of follow up :Day 28 for the primary endpoint

DETAILED DESCRIPTION:
Secondary (exploratory) objectives

* To evaluate the impact of 300mL convP on mortality
* To evaluate the impact of 300mL convP on hospital admission
* To evaluate the impact of 300mL convP on admission to ICU
* To evaluate the impact of 300mL convP on duration of symptoms
* To evaluate the impact of 300mL convP in relation to the age and clinical frailty of the patient

ELIGIBILITY:
Inclusion Criteria:

* RT-PCR-confirmed COVID-19.
* Symptomatic (e.g but not limited to fatigue, fever, cough, dyspnoea, loss of taste or smell, diarrhea, falls or confusion)
* 70 years or older OR 50-69 years and 1 or more of the risk factors described in the protocol

Exclusion Criteria:

* Life expectancy <28 days in the opinion of the treating physician
* Patient or legal representative is unable to provide written informed consent
* Symptomatic for 8 days or more
* Being admitted to the hospital at the informed consent procedure
* Known previous history of transfusion-related acute lung injury
* Known Immunoglobulin A (IgA) deficiency

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Highest disease status | 28 days following transfusion of convP or FFP
  Highest disease status on the 5-point ordinal disease severity scale in the convP group will be compared with the FFP group.

SECONDARY OUTCOMES:
Percentage of deaths | 28 days following transfusion of convP or FFP
  Percentage of deaths in the convP group compared to the FFP group
Percentage of hospital admissions | 28 days following transfusion of convP or FFP
  Percentage of hospital admissions in the convP group compared to the FFP group
Percentage of ICU admissions | 28 days following transfusion of convP or FFP
  Percentage of ICU admissions in the convP group compared to the FFP group
Disease duration in days of symptoms | 28 days following transfusion of convP or FFP
  Disease duration in days of symptoms in the convP group compared to the FFP group
Age and clinical frailty score | 28 days following transfusion of convP or FFP
  Age and clinical frailty score stratified analysis of percentage of primary endpoint following transfusion of convP versus FFP.

OTHER OUTCOMES:
Highest disease status stratified by presence of neutralizing antibodies and by symptom duration at baseline | 28 days following transfusion of convP or FFP
  Analysis of primary endpoint following transfusion of convP versus FFP stratified by the presence of neutralizing antibodies at baseline and by symptom duration at baseline.
Change in proportion of detectable SARS-Cov-2 RT-PCR results | Day 3, 7, 14 and 28 following transfusion of convP or FFP
  Change in proportion of detectable SARS-CoV-2 RT-PCR results at day 3, 7, 14 and 28 following transfusion according to the presence of neutralizing antibodies at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bart Rijnders, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (11):
- Netherlands (11):
  - Erasmus Medical Center, Rotterdam, South Holland
  - Meander Medisch Centrum, Amersfoort
  - Rijnstate Ziekenhuis, Arnhem
  - Amphia Ziekenhuis, Breda
  - Groene Hart Ziekenhuis, Gouda
  - University Medical Center Groningen (UMCG), Groningen
  - Spaarne Gasthuis, Haarlem
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leids Universitair Medisch Centrum, Leiden
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Bernhoven Hospital, Uden

REFERENCES:
- [Derived] Millat-Martinez P, Gharbharan A, Alemany A, Rokx C, Geurtsvankessel C, Papageorgiou G, van Geloven N, Jordans C, Groeneveld G, Swaneveld F, van der Schoot E, Corbacho-Monne M, Ouchi D, Piccolo Ferreira F, Malchair P, Videla S, Garcia Garcia V, Ruiz-Comellas A, Ramirez-Morros A, Rodriguez Codina J, Amado Simon R, Grifols JR, Blanco J, Blanco I, Ara J, Bassat Q, Clotet B, Baro B, Troxel A, Zwaginga JJ, Mitja O, Rijnders BJA; CoV-Early study group; COnV-ert study group. Prospective individual patient data meta-analysis of two randomized trials on convalescent plasma for COVID-19 outpatients. Nat Commun. 2022 May 11;13(1):2583. doi: 10.1038/s41467-022-29911-3. PMID 35546145